CLINICAL TRIAL: NCT06661421
Title: Effects of Dry Needling on Spasticity, Range of Motion, and Functional Mobility Among Children With Cerebral Palsy
Brief Title: Effects Of Dry Needling On Mobility Among Children With Cerebral Palsy
Acronym: DRYSPARC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0701
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Palsy (CP); Spasticity; Range of Motion; Functional Mobility
Keywords: Cerebral Palsy; Spasticity; Dry Needling; Range of Motion; Functional Mobility
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Dry Needling

STUDY DESIGN:
Intervention Model Description: A sample size of 38 was calculated using Epitool online software, and the mean values of dynamic balance from the previous study were taken. By adding a 10% attrition rate (34+4), the sample size will be 38.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols, and possible efforts will be put to mask both groups about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dry Needling Group (Experimental): Group A will receive Dry Needling Therapy (DNT) along with routine physical therapy. Each session includes a 5-minute warm-up, stretching, and strengthening exercises. Hamstring stretches will be done with the child supine, one leg flat, and the opposite hip flexed to 90°. Active knee extension will be held for 5 seconds, followed by a 40-second assisted stretch, repeated five times. If a short psoas is detected, psoas stretching will be done prone, with assisted hip extension for 5 seconds and a 40-second hold, repeated five times. Strengthening exercises, including squats, heel rises, and step-ups with a loaded backpack, will target the lower extremities. The program lasts one month with three sessions per week, gradually increasing in intensity. Dry Needling (DN) uses 0.30 × 50 mm needles, applying the fast-in, fast-out technique for 1 minute per muscle. DN is done once per week for 10 weeks, with at least 48 hours between treatments.
  Interventions: Device: Dry Needling
- Conventional Therapy Group (Other): Sessions will include a 5-minute warm-up, stretching, and strengthening exercises. Hamstring stretches will be done with the child supine, one leg flat, and the opposite hip flexed to 90°. Active knee extension will be held for 5 seconds, followed by a 40-second assisted stretch, repeated five times. If a short psoas is detected, a prone psoas stretch will involve assisted hip extension for 5 seconds, followed by a 40-second hold, repeated five times. Strengthening exercises like squats, heel raises, and step-ups with a loaded backpack will target the lower extremities. The program will last one month, with three weekly sessions focusing on hamstring stretches and progressive resistance exercises.
  Interventions: Other: Cerebral Palsy conventional Treatment

INTERVENTIONS:
Device: Dry Needling — This intervention combines Dry Needling Therapy (DNT) with routine physical therapy for children with spastic cerebral palsy. The experimental group will receive DNT alongside physical therapy, while the control group will undergo only physical therapy. Routine Physical Therapy includes a warm-up, stretching, and strengthening exercises like hamstring stretches and squats, adjusted over a month with increasing intensity. Dry Needling targets the gastrocnemius muscle using a fast-in, fast-out technique with sterile needles, applied weekly for 10 weeks. This combined approach aims to reduce spasticity, improve mobility, and enhance range of motion, distinguishing it from standard therapies.
  Arms: Dry Needling Group
Other: Cerebral Palsy conventional Treatment — Sessions will include a 5-minute warm-up, stretching, and strengthening exercises. Hamstring stretches will be done with the child supine, one leg flat, and the opposite hip flexed to 90°. Active knee extension will be held for 5 seconds, followed by a 40-second assisted stretch, repeated five times. If a short psoas is detected, a prone psoas stretch will involve assisted hip extension for 5 seconds, followed by a 40-second hold, repeated five times. Strengthening exercises like squats, heel rises, and step-ups with a loaded backpack will target the lower extremities. The program will last one month, with three sessions per week, focusing on hamstring stretches and progressive resistance exercises.
  Arms: Conventional Therapy Group

SUMMARY:
This study explores the potential of dry needling as a treatment for spasticity in the foot among children with cerebral palsy (CP). Dry needling involves inserting fine needles into specific trigger points or tight muscles without injecting any substances, aiming to relieve pain, improve muscle function, and promote tissue healing. In CP-related foot spasticity, dry needling may target hypertonic muscles, inducing a local twitch response that helps release muscle tension, reduce spasticity, and enhance overall muscle function. The technique may also stimulate sensory nerves and trigger the release of endorphins, contributing to pain relief and muscle relaxation.

While dry needling has shown effectiveness in reducing spasticity and improving muscle function in adults with conditions such as post-stroke, there is limited research on its benefits for children with CP. This randomized controlled trial aims to address this gap by evaluating the impact of dry needling on spasticity, range of motion, and functional mobility in children with CP.

DETAILED DESCRIPTION:
The study will be conducted at Bliss Center of Care and Therapy in Faisalabad, involving 38 participants aged 6 to 12 years, all diagnosed with spastic cerebral palsy and classified under the Gross Motor Function Classification System (GMFCS) levels I-II. Participants will be divided into two groups: an experimental group receiving dry needling therapy (DNT) and routine physical therapy (RPT) and a control group receiving RPT only. Critical exclusion criteria include recent interventions, bleeding disorders, fixed joint deformities, recent seizures, Botulinum Toxin injections, or contraindications to dry needling.

Outcomes will be measured using the Wartenberg Pendulum Test, Active and Passive Ankle Dorsiflexion Range of Motion, and the Timed Up and Go Test, which will be assessed before and after a 10-week intervention. Data will be analyzed using SPSS version 23.0 to determine the efficacy of dry needling in managing spasticity in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* Age: 6 to 12 years old
* Walking ability at Gross Motor Function Classification System levels I to II
* Modified Modified Ashworth Scale (MAS) score higher than equal to 1 (score up to 2)
* Ability to understand and execute orders
* No ongoing rehabilitation intervention

Exclusion Criteria:

* Recent introduction of a new intervention in addition to previous treatments
* Presence of bleeding disorders or skin conditions
* Skin sensitivity issues
* History of seizures within the past six months
* Previous administration of BTX-A injection within the last 6 months
* Presence of
* contraindications to dry needling
* Lack of consent to participate in the study

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2024-09-24 (Actual); Primary Completion 2024-12-15 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Wartenberg Pendulum Test | The Wartenberg Pendulum Test will be conducted once upon the start of the trial (Pre-test) and once at the end of trial (Post-Test) to check the effect of the research. In total, the Wartenberg Pendulum Test will be performed two times.
  In the Wartenberg Pendulum Test, the extended leg of a supine individual is allowed to fall freely, and under normal circumstances, it swings back and forth like a pendulum. However, in spastic limbs, the viscoelastic properties and heightened stretch reflexes dampen the swing, limiting its motion. To conduct the test, the individual should be seated with legs hanging freely and their back supported. They must fully relax the muscles, especially in the tested leg, with gentle support under the thigh if needed. The examiner holds the lower leg above the ankle, ensuring the knee is straight but not hyperextended, and then gently moves the leg to the side before releasing it to swing freely. The examiner observes the initial swing amplitude and subsequent swings, noting any decrease and counting swings until rest. The test is repeated on the other leg for comparison. Reduced amplitude or asymmetry suggests spasticity and the relaxation index (R2 ratio) is commonly measured.

SECONDARY OUTCOMES:
Ankle Dorsiflexion Range of Motion | The Ankle dorsiflexion ROM will be conducted once upon the start of the trial (Pre-test) and once at the end of trial (Post-Test) to check the effect of the research. In total, the Ankle dorsiflexion ROM will be performed two times.
  Ankle dorsiflexion ROM, active and passive, is assessed with the patient supine and the knee extended, using a manual goniometer. The fulcrum is placed on the lateral malleolus, the stationary arm aligned with the fibula, and the movable arm parallel to the fifth metatarsal. Test-retest reliability of ankle dorsiflexion ROM using a universal goniometer has shown ICC values ranging from 0.75 to 0.96, with a comprehensive score of 0.91, indicating excellent reliability.
The Ankle dorsiflexion ROM will be conducted upon the start of the trial (Pre-test) and once at the end of trial (Post-Test) to check the effect of the research. In total, the Ankle dorsiflexion ROM will be performed two times. | The Modified Timed Up and Go Test will be conducted once at the start of the trial (Pre-test) and once at the end of trial (Post-Test) to check the effect of the research. In total, the Modified Timed Up and Go will be performed two times.
  The Modified Timed Up and Go (TUG) test evaluates functional ambulatory mobility and dynamic balance in children. It measures the time a child takes to stand seated, walk 3 meters, touch a star on the wall, return to the chair, and sit down. For the procedure, the child starts by sitting on a stool with their feet flat on the floor, knees, and hips at 90° flexion. They are then instructed to stand, walk 3 meters, touch the star on the wall, return to the chair, and sit down. The child may wear regular footwear or orthoses, and walking aids are permitted, but no physical assistance is provided. The timing is recorded with a stopwatch, and there is no time limit; the child may rest if needed without sitting down. The Modified TUG test demonstrates excellent reliability, with an intraclass correlation coefficient (ICC) of 0.99 for both within-session and test-retest assessments, making it a valuable tool for evaluating mobility in pediatric rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Maheen Ahmad Khan, MS*, Principal Investigator — Riphah International Univerisity
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ghannadi S, Shariat A, Ansari NN, Tavakol Z, Honarpishe R, Dommerholt J, Noormohammadpour P, Ingle L. The Effect of Dry Needling on Lower Limb Dysfunction in Poststroke Survivors. J Stroke Cerebrovasc Dis. 2020 Jun;29(6):104814. doi: 10.1016/j.jstrokecerebrovasdis.2020.104814. Epub 2020 Apr 21. PMID 32327366
- [Background] Cruz-Montecinos C, Nunez-Cortes R, Bruna-Melo T, Tapia C, Becerra P, Pavez N, Perez-Alenda S. Dry needling technique decreases spasticity and improves general functioning in incomplete spinal cord injury: A case report. J Spinal Cord Med. 2020 May;43(3):414-418. doi: 10.1080/10790268.2018.1533316. Epub 2018 Oct 22. PMID 30346254